CLINICAL TRIAL: NCT00456352
Title: Phase IV Study of Duodenal Exclusion for the Treatment of Type 2 Diabetes Mellitus (T2DM)
Brief Title: Duodenal Exclusion for the Treatment of T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS07004
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Procedure: duodenal exclusion

SUMMARY:
Evaluation of duodenal exclusion procedure for the treatment of T2DM

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 65 years
2. BMI between 23 and 34
3. Oral agents or insulin to control T2DM
4. Inadequate control of diabetes as defined as HbA1c >/ 7.5
5. Understanding of the mechanisms of action of the treatment

Exclusion Criteria:

1. More than 10 years of T2DM diagnosis
2. More than 7 years of insulin use
3. Previous abdominal operations
4. Coagulopathy
5. Liver cirrhosis
6. Unable to comply with study requirements, follow-up schedule or give valid consent.
7. Currently pregnant.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Treatment success based on patients' glycemic control. | 2 weeks, 3 months, 6 months, 9 months, 12 months

SECONDARY OUTCOMES:
Physiologic measurements, Comorbidity improvement, Improvement in QOL. | 2 weeks, 3 months, 6 months, 9 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Noreen A Gannon, Study Director — Medtronic - MITG; Ricardo Cohen, MD, Principal Investigator — Hospital São Camilo
Locations (1):
- Hospital São Camilo, São Paulo, Brazil